CLINICAL TRIAL: NCT04153721
Title: Evaluation of a Digital Perioperative Support Solution for Colorectal Surgery: Compliance and Impact on Patients
Brief Title: Impact Study of a Digital Solution for Patient Engagement
Acronym: Get Ready
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IHU Strasbourg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-007
Record Dates: First submitted 2019-10-21; First posted 2019-11-06 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Cancer
Keywords: enhanced recovery; rehabilitation; prehabilitation; patient engagement; digital health; e-health; colorectal surgery; preparation; follow-up; patient empowerment
MeSH Terms: conditions — Colorectal Neoplasms; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Digital Solution (Experimental): The proposed digital solution aims to improve the patient's preparation for his colorectal surgery and follow his rehabilitation after surgery, by reinforcing his compliance with existing protocols and enriching it with complementary practices
  Interventions: Behavioral: Name Digital Solution

INTERVENTIONS:
Behavioral: Name Digital Solution — The digital solution offers a pre-operative program of information (pathology, treatment modalities, protocols to be followed) and training (stress management, psychological support, optional: nutritional preparation, physical exercise, reduction of alcohol and tobacco consumption).
  In the post-operative phase, patients must daily assess their state of health (temperature, weight, wound, nausea / vomiting, urine / stool) and well-being (physical, moral, sleep, pain), from day 1 to day 7 after discharge, to facilitate the detection of complications by the medical team

SUMMARY:
The Institute of Image-Guided Surgery (IHU) of Strasbourg develops new minimally invasive therapies, the benefit of which is maximized by an integrated approach to the care pathway (pre, per and postoperative).

Encouraging patient engagement in the process responds to its growing demand for information and consideration, enhances its care experience and clinical outcomes.

Medtronic has designed an digital solution for patient engagement (current name: "Get Ready") for scheduled colorectal surgery. The IHU is a pilot experiment site for this solution. This research protocol, of which the IHU is the promoter, aims at evaluating the use and the impact of this solution made available to the patients of the Hepato-Digestive Pole (PHD) of the New Civil Hospital.

The solution deployed at the Strasbourg IHU aims to improve the patient's preparation for his colorectal surgery and follow his rehabilitation after surgery, by reinforcing his compliance with existing protocols and enriching it with complementary practices.

The solution is not a medical device. It is limited to advice, monitoring and restitution of data declared by the patient; it is not intended to prevent, diagnose or treat the pathology; it is independent of any other medical device.

This study aims to assess the pre-operative impact of the solution, in terms of patients' adherence to the pre-operative program and correlations with their physical and psychological condition until their admission to surgery. The secondary purpose of the study is to precise the acceptability of the solution.

DETAILED DESCRIPTION:
The Institute of Image-Guided Surgery (IHU) of Strasbourg develops new minimally invasive therapies, the benefit of which is maximized by an integrated approach to the care pathway (pre, per and postoperative).

Encouraging patient engagement in the process responds to its growing demand for information and consideration, enhances its care experience and clinical outcomes. Patient engagement promotes accelerated rehabilitation and reduces complications and readmissions, which is also beneficial in terms of public health.

Medtronic has designed a digital solution for patient engagement (current name: "Get Ready") for scheduled colorectal surgery, for which the IHU is a pilot experiment site. This research protocol aims at evaluating the use and the impact of this solution made available to the patients of the Hepato-Digestive Pole (PHD) of the New Civil Hospital.

Multiple professionals dispense instructions and information to patients. The active accompaniment of the patient in his rehabilitation process is carried out mainly in the postoperative phase, during the hospital stay.

The solution deployed at the Strasbourg IHU aims to improve the patient's preparation for his colorectal surgery and follow his rehabilitation after surgery, by reinforcing his compliance with existing protocols and enriching it with complementary practices.

The solution offers a pre-operative program of information (pathology, treatment modalities, protocols to be followed) and training (stress management, psychological support, optional: nutritional preparation, physical exercise, reduction of alcohol and tobacco consumption). In the post-operative phase, patients must daily assess their state of health (temperature, weight, wound, nausea / vomiting, urine / stool) and well-being (physical, moral, sleep, pain), from day 1 to day 7 after discharge, to facilitate the detection of complications by the medical team.

The program is personalized by patient, according to its management (type of surgery, duration of the program) and its state of health (choice of options adapted by the doctor).

The solution has three components to interact with the patient:

* A website, offering information and activities adapted to the patient's journey. A second site allows the licensed care team to track adherence and patient-reported data.
* SMS (Short Message Service) notifications, for the patient who can and wants to receive SMS. It encourages the monitoring of the program (reminders).
* An on-site IHU support team, accessible by phone and email. She ensures the smooth running of the program, supervises the information declared by the patient and relays his questions to the relevant interlocutors (care team, technical experts).

The solution is not a medical device. It is limited to advice, monitoring and restitution of data declared by the patient; it is not intended to prevent, diagnose or treat the pathology; it is independent of any other medical device.

The solution processes personal information. Particular vigilance is therefore given to security: compliance with legislation, state-of-the-art techniques used, respect for privacy from the upstream and by default, transparency and control, security measures (eg data encryption, double authentication, lack of interfaces to other information systems, accredited health host).

According to the literature, the preparation of the patient for surgery makes it possible to shorten the length of stay, the perioperative morbidity, the delay to come back to normal activity. This medical impact results in a reduction in post-operative costs (reduction of the length of stay, complications and readmissions), for the health facility and the payer. Improvement and systematization of the solution should help generate these savings.

The impact of the solution on the workload and the organization of the care team is to be specified.

This study aims to assess the pre-operative impact of the solution, in terms of patients' adherence to the pre-operative program and correlations with their physical and psychological condition until their admission to surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Major patient candidate for a scheduled colorectal surgery and whose admission is expected within 8 days minimum
2. Patient with an email address and an internet connection
3. Patient able to receive and understand information about the study and give written informed consent

Exclusion Criteria:

1. Patient under the age of 18 years old.
2. Pregnant or lactating patient
3. Patient in exclusion period (determined by a previous or a current study)
4. Patient under guardianship, trusteeship or the protection of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Evaluation, during the preoperative phase, of patients' compliance to the program, assessed by a completeness rate. | From the inclusion to the surgery
  Positive correlations between compliance and improvement of the patient's condition will help demonstrate the value of the solution. The first part of the primary endpoint of the study is the average rate of completeness of the preoperative program: percentage based on the status (done / not done) of pre-operative tasks specific to each patient
Change, during the preoperative phase, of the physical condition of the patients, assessed by 6MTW scoring. | At the start of the program (6 weeks before the surgery) and at the admission before the surgery
  Positive correlations between compliance and improvement of the patient's condition will help demonstrate the value of the solution. The second part of the primary endpoint of the study is the correlation between the patient compliance and the evolution of the physical condition :
  comparison between two walk tests, one done at the inclusion, the other when admitted for surgery. The result of the walk test is the distance travelled in meters during the test (6 minutes) by the patient.
Change, during the preoperative phase, of the psychological condition of the patients, assessed by the PHQ8 questionnaire scoring. | At the start of the program (6 weeks before the surgery) and at the admission before the surgery
  Positive correlations between compliance and improvement of the patient's condition will help demonstrate the value of the solution. The third part of the primary endpoint of the study is the correlation between the patient compliance and the evolution of the psychological condition assessed by the questionnaire PHQ8 (Brief "Patient Health Questionnaire" depression scale): questions the existence and intensity of depressive symptoms (score from 0 to 24 in case of severe depression).
Change, during the preoperative phase, of the psychological condition of the patients, assessed by GAD7 questionnaire scoring. | At the start of the program (6 weeks before the surgery) and at the admission before the surgery
  Positive correlations between compliance and improvement of the patient's condition will help demonstrate the value of the solution. The fourth part of the primary endpoint of the study is the correlation between the patient compliance and the evolution of the psychological condition evaluated by the questionnaire GAD7 ("Generalized Anxiety Disorder 7"-item): indicates the severity of the anxiety (score from 0 to 21 in case of generalized anxiety disorder)

SECONDARY OUTCOMES:
Evaluation of patients' compliance with their post-operative program | Everyday for 7 days after the discharge from hospital and on the 14th day after the discharge from hospital
  Completeness rate of the postoperative program. This rate is calculated according to the status (done or not done) of the tasks to be performed by the patient after the surgical procedure: daily evaluations the first week and the 14th day after discharge from hospital. Task status is plotted in the digital solution.
Persistence of program compliance between pre- and post-operative phases | From the inclusion to the end of participation
  Persistence of the program compliance, defined as the difference between the pre and the postoperative completeness rate of the program
Patient satisfaction regarding the program | 2 days before the surgery and on the 14th day after the discharge from hospital
  The satisfaction is assessed on all patients by three questions (useful, adapted, promotable program). The scores obtained on these three questions will be measured pre-operatively, post-operatively and averaged over the whole program. These scores are calculated automatically by the solution.
Evaluation, during the preoperative phase, of patient use of the program without compliance, assessed by a rate of undone activities | from 6 weeks before the surgery up to the surgery
  For patients with a preoperative physical activity and/or nutritional program prescribed, number of declared as undone activities compared to the total number of prescribed activities
Patient interactions with the help desk of the solution | from the inclusion to the end of participation
  Rate of patient interactions with the help desk of the solution, defined as the mean number of phone call and emails per patient
Evaluation of the solution and its use by the patient | Visit Day 30
  Qualitative interview with the patient, carried out during his follow-up consultation J30
Evaluation of the solution and its use by health care providers | End of study
  Qualitative interview with health care providers (physicians, interns), carried out at the end of the study
Evaluation of the postoperative complication rate | Visit Day 30
  Number of postoperative complications identified 30 days after the surgery
Evaluation of duration of hospital stays | from the day before the admission until the end of hospitalisation
  Quantification of the hospital stay duration, defined as defined by the difference between the date of discharge from hospital and the date of admission
Evaluation of the number of postoperative critical values | 7 days after the discharge of the hospital
  The number of post-operative critical values detected following daily assessments in the week following discharge from hospital, in accordance with the thresholds defined by the care team

CONTACTS AND LOCATIONS:
Overall Officials: Didier Mutter, MD, PhD, Principal Investigator — Service Chirurgie Digestive et Endocrinienne, Nouvel Hôpital Civil de Strasbourg
Locations (1):
- Service de Chirurgie Digestive et Endocrinienne, NHC, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Santa Mina D, Clarke H, Ritvo P, Leung YW, Matthew AG, Katz J, Trachtenberg J, Alibhai SM. Effect of total-body prehabilitation on postoperative outcomes: a systematic review and meta-analysis. Physiotherapy. 2014 Sep;100(3):196-207. doi: 10.1016/j.physio.2013.08.008. Epub 2013 Nov 13. PMID 24439570
- [Background] Wind J, Polle SW, Fung Kon Jin PH, Dejong CH, von Meyenfeldt MF, Ubbink DT, Gouma DJ, Bemelman WA; Laparoscopy and/or Fast Track Multimodal Management Versus Standard Care (LAFA) Study Group; Enhanced Recovery after Surgery (ERAS) Group. Systematic review of enhanced recovery programmes in colonic surgery. Br J Surg. 2006 Jul;93(7):800-9. doi: 10.1002/bjs.5384. PMID 16775831
- [Background] Wang L, Lee M, Zhang Z, Moodie J, Cheng D, Martin J. Does preoperative rehabilitation for patients planning to undergo joint replacement surgery improve outcomes? A systematic review and meta-analysis of randomised controlled trials. BMJ Open. 2016 Feb 2;6(2):e009857. doi: 10.1136/bmjopen-2015-009857. PMID 26839013
- [Background] Li C, Carli F, Lee L, Charlebois P, Stein B, Liberman AS, Kaneva P, Augustin B, Wongyingsinn M, Gamsa A, Kim DJ, Vassiliou MC, Feldman LS. Impact of a trimodal prehabilitation program on functional recovery after colorectal cancer surgery: a pilot study. Surg Endosc. 2013 Apr;27(4):1072-82. doi: 10.1007/s00464-012-2560-5. Epub 2012 Oct 9. PMID 23052535
- [Background] van der Meij E, Anema JR, Leclercq WKG, Bongers MY, Consten ECJ, Schraffordt Koops SE, van de Ven PM, Terwee CB, van Dongen JM, Schaafsma FG, Meijerink WJHJ, Bonjer HJ, Huirne JAF. Personalised perioperative care by e-health after intermediate-grade abdominal surgery: a multicentre, single-blind, randomised, placebo-controlled trial. Lancet. 2018 Jul 7;392(10141):51-59. doi: 10.1016/S0140-6736(18)31113-9. Epub 2018 Jun 21. PMID 29937195
- [Background] Mayo NE, Feldman L, Scott S, Zavorsky G, Kim DJ, Charlebois P, Stein B, Carli F. Impact of preoperative change in physical function on postoperative recovery: argument supporting prehabilitation for colorectal surgery. Surgery. 2011 Sep;150(3):505-14. doi: 10.1016/j.surg.2011.07.045. PMID 21878237
- [Background] Snow R, Granata J, Ruhil AV, Vogel K, McShane M, Wasielewski R. Associations between preoperative physical therapy and post-acute care utilization patterns and cost in total joint replacement. J Bone Joint Surg Am. 2014 Oct 1;96(19):e165. doi: 10.2106/JBJS.M.01285. PMID 25274793
- [Background] van Rooijen S, Carli F, Dalton S, Thomas G, Bojesen R, Le Guen M, Barizien N, Awasthi R, Minnella E, Beijer S, Martinez-Palli G, van Lieshout R, Gogenur I, Feo C, Johansen C, Scheede-Bergdahl C, Roumen R, Schep G, Slooter G. Multimodal prehabilitation in colorectal cancer patients to improve functional capacity and reduce postoperative complications: the first international randomized controlled trial for multimodal prehabilitation. BMC Cancer. 2019 Jan 22;19(1):98. doi: 10.1186/s12885-018-5232-6. PMID 30670009
- [Background] Lin LY, Wang RH. Abdominal surgery, pain and anxiety: preoperative nursing intervention. J Adv Nurs. 2005 Aug;51(3):252-60. doi: 10.1111/j.1365-2648.2005.03502.x. PMID 16033593
- [Background] Adamina M, Kehlet H, Tomlinson GA, Senagore AJ, Delaney CP. Enhanced recovery pathways optimize health outcomes and resource utilization: a meta-analysis of randomized controlled trials in colorectal surgery. Surgery. 2011 Jun;149(6):830-40. doi: 10.1016/j.surg.2010.11.003. Epub 2011 Jan 14. PMID 21236454
- [Background] Pecorelli N, Fiore JF Jr, Gillis C, Awasthi R, Mappin-Kasirer B, Niculiseanu P, Fried GM, Carli F, Feldman LS. The six-minute walk test as a measure of postoperative recovery after colorectal resection: further examination of its measurement properties. Surg Endosc. 2016 Jun;30(6):2199-206. doi: 10.1007/s00464-015-4478-1. Epub 2015 Aug 27. PMID 26310528
- [Background] Hijazi Y, Gondal U, Aziz O. A systematic review of prehabilitation programs in abdominal cancer surgery. Int J Surg. 2017 Mar;39:156-162. doi: 10.1016/j.ijsu.2017.01.111. Epub 2017 Feb 2. PMID 28161527
- [Background] Inoue T, Ito S, Kanda M, Niwa Y, Nagaya M, Nishida Y, Hasegawa Y, Koike M, Kodera Y. Preoperative six-minute walk distance as a predictor of postoperative complication in patients with esophageal cancer. Dis Esophagus. 2020 Mar 5;33(2):doz050. doi: 10.1093/dote/doz050. PMID 31111872
- [Background] Chen YC, Chen KC, Lu LH, Wu YL, Lai TJ, Wang CH. Validating the 6-minute walk test as an indicator of recovery in patients undergoing cardiac surgery: A prospective cohort study. Medicine (Baltimore). 2018 Oct;97(42):e12925. doi: 10.1097/MD.0000000000012925. PMID 30335028
- [Background] Marek W, Marek E, Vogel P, Muckenhoff K, Kotschy-Lang N. [A new procedure for the estimation of physical fitness of patients during clinical rehabilitation using the 6-minute-walk-test]. Pneumologie. 2008 Nov;62(11):643-54. doi: 10.1055/s-2008-1038204. Epub 2008 Aug 18. German. PMID 18711694
- [Background] Kroenke K, Strine TW, Spitzer RL, Williams JB, Berry JT, Mokdad AH. The PHQ-8 as a measure of current depression in the general population. J Affect Disord. 2009 Apr;114(1-3):163-73. doi: 10.1016/j.jad.2008.06.026. Epub 2008 Aug 27. PMID 18752852
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- See also: French National Authority for Health, Recommendation of good practice: Adult characterized depressive episode : primary care. October 2017 — https://www.has-sante.fr/jcms/c_1739917/fr/episode-depressif-caracterise-de-l-adulte-prise-en-charge-en-premier-recours